CLINICAL TRIAL: NCT04489745
Title: Stereotactic Body Radiotherapy (SBRT) for Localized Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VALosAngeles
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT and ADT (Experimental): Patients undergo SBRT to a dose of 40 Gy in 5 fractions to prostate, and optional 25 Gy in 5 fractions to SVs and Pelvic LNs, with 9 months of Androgen Deprivation Therapy
  Interventions: Radiation: SBRT; Drug: Androgen deprivation therapy (ADT)

INTERVENTIONS:
Radiation: SBRT
Drug: Androgen deprivation therapy (ADT)

SUMMARY:
This is a trial of 5 fraction SBRT combined with androgen deprivation therapy for patients with localized high-risk or unfavorable intermediate risk prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary non-metastatic adenocarcinoma of the prostate
* High-risk or unfavorable intermediate-risk as defined below:

High-risk localized prostate cancer, as defined by any one of the following factors:

Pre-biopsy or any PSA ≥20 prior to enrollment, or Gleason score 8 or higher on any biopsy core, or cT3a or higher.

Unfavorable intermediate risk localized prostate cancer, as defined as any of the following factors:

Gleason score of 4+3 or higher on any biopsy core, or Gleason score 3+4 and >50% biopsy cores positive, or The presence of any two of the following: PSA>10, cT2b-c, Gleason score 3+4 in any core

* No pelvic nodal metastases (based on CT or MRI findings)
* No distant metastases, based upon:

CT scan or MRI of the pelvis within 120 days prior to registration, Bone scan within 120 days prior to registration; if the bone scan is suspicious, a plain x-ray and/or MRI must be obtained to rule out metastasis

* Age ≥ 18
* KPS ≥ 70 (or ECOG 0-2)
* Ability to understand, and willingness to sign, the written informed consent

Exclusion Criteria:

* Patients with low-risk or favorable intermediate-risk prostate cancer do not meet inclusion criteria (these patients would be eligible for SBRT off-trial as a standard of care option)
* Patients with any evidence of distant metastases
* Hormonal therapy (LHRH agonist or oral anti-androgen) exceeding 7 months prior to registration
* Prior cryosurgery, HIFU or brachytherapy of the prostate
* Prior pelvic radiotherapy
* History of Crohn's Disease or Ulcerative Colitis

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 5 years
  progression is defined by biochemical (phoenix definition), clinical, or radiographic

IPD SHARING:
Plan to Share IPD: Undecided